CLINICAL TRIAL: NCT05272436
Title: Home-based Immersive Virtual Reality Physical Rehabilitation in Paediatric Patients for Upper Limb Motor Impairment
Brief Title: Using Virtual Reality for Rehabilitation of Upper Limbs at Home Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AA14673868
Record Dates: First submitted 2022-02-25; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Upper Limb Injury; Virtual Reality; Rehabilitation; Paediatric
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Intervention Model Description: This study aimed to explore:
  * patients, clinicians, family members perceptions of the effect of IVR on ULMI rehabilitation (range of movement (ROM) recovery)
  * patient perceptions of the usability, quality of live, acceptability, engagement with and enjoyment of IVR scenarios;
  * occupational therapies perceptions about the usability and implications of the IVR technology within a patient rehabilitation at home.
  Methods: This was a small-scale mixed methods (quantitative and qualitative) study.
  Patients: paediatric patients recruited from Sheffield Children's Foundation Hospital Trust in England, UK, their parents, and an occupational therapist (OT) from the Sheffield Children's Foundation Hospital Trust for Burns, Plastics, and Orthopaedics participated in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients IVR for Upper Limb Motor Impairment Rehabilitation in children and at home trial (Experimental): For the purpose of the trial, patients had their usual OT/PT appointments but were asked to use the IVR games to do the prescribed home exercises. Before consenting to participate, each patient was offered a 5-10 minute experience of the game to familiarise themselves with how it worked and to check for problems. Written and verbal consents were taken from parents and children.
  The pre-trial PedsQL was administered in the initial OT/PT appointment. Children were then asked to use the IVR system for approximately 15 minutes twice a day. Trial participation lasted three weeks during the prescribed treatment weeks.
  Following the at-home trial, patients and parents returned the equipment to the clinic in the final appointment and the SUS and the post-trial Peds QL were administrated by OT/PT in person. In addition, they participated in semi-structured interviews as described above.
  Interventions: Device: Virtual Reality Upper Limb Motor Impairment Rehabilitation
- Occupational Therapist perceptions of the effectiveness of the IVR (Other): She recruited the patients, gave out devices, administered the outcome measures and provided us with feedback about their experience with the VR game.
  At the end of the trial, an interview (10 minutes) with the OT was conducted by a research nurse.
  Interventions: Device: Virtual Reality Upper Limb Motor Impairment Rehabilitation

INTERVENTIONS:
Device: Virtual Reality Upper Limb Motor Impairment Rehabilitation — Patients wore a VR headset while undergoing their physical rehabilitation at home
  Other Names: No intervention

SUMMARY:
The IVR games have been enhanced to include more levels. The new aspects to be tested in this study are new IVR exercises that would be made upper limb rehab designed for children for home use, as repeated sessions with progression through different levels could improve the prospect of good functional recovery. A new wireless headset has recently become available, which will enable the IVR to be run without the need for separate equipment, thereby making home use possible as no complicated set-up will be required.

This project aims to explore the feasibility, acceptability and perceived effectiveness of an improved suite of Immersive Virtual Reality (IVR) system suitable for Upper Limb Motor Impairment (ULMI) rehabilitation for children at home. A multidirectional perspective has been adopted, including patients, caregivers, and clinical staff.

The aims and objectives of the clinical feasibility trial are:

* to investigate the potential of IVR for ULMI rehabilitation (range of motion recovery) at home compared to usual physical therapy in a small sample of paediatric patients.
* to measure the impact of the interventions from a mixed methods (quantitative and qualitative) and a multidirectional perspective (patients, clinicians, family members).

DETAILED DESCRIPTION:
This project builds upon a previous MRC 'Confidence in Concept' feasibility project which developed Virtual Reality (VR) games for participants at Sheffield Children's Hospital to do arm rehabilitation movements such that they become so engrossed in the IVR they become much less aware of any pain or discomfort linked to the exercises.

Patients (and carer where appropriate) would be involved in the design of the scenarios, the protocol, patient information sheets, and the project steering group. Research nurses will download anonymised usage data from the VR headset used at home and interview participants. All data will feed into an evaluation which will demonstrate the concept and acceptability of using IVR at home.

Procedure Patients usually have a 20-30 minutes appointment during which the OT/PT reviews their previously prescribed home exercise regime with them, measures ROM, and explains and discusses new home exercises. For the purpose of the trial, patients had their usual OT/PT appointments but were asked to use the IVR games to do the prescribed home exercises. Before consenting to participate, each patient was offered a 5-10 minute experience of the game to familiarise themselves with how it worked and to check for problems. Written and verbal consents were taken from parents and children.

The pre-trial PedsQL was administered in the initial OT/PT appointment. Children were then asked to use the IVR system for approximately 15 minutes twice a day. Trial participation lasted three weeks during the prescribed treatment weeks.

Following the at-home trial, patients and parents returned the equipment to the clinic in the final appointment and the SUS and the post-trial Peds QL were administrated by OT/PT in person. In addition, they participated in semi-structured interviews as described above.

At the end of the trial, an interview (10 minutes) with the OT was conducted by a research nurse.

ELIGIBILITY:
Inclusion Criteria:

* aged 7-16
* upper limb injuries, for which they are receiving rehabilitative care
* able to speak and understand English.

Exclusion Criteria:

1. injuries to the face or head that could hinder the correct positioning of the headset or pose an infection risk;
2. A learning impairment that could hinder the understanding of the task;
3. A history of severe motion sickness;
4. Mental health problems;
5. Inability to speak and understand English.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Ratings of child participant's movement during physiotherapy sessions: Goniometer (Standard BASELINE® 12-inch) | Three weeks
  Goniometer device (Standard BASELINE® 12-inch plastic goniometer, (Model 12-1000-Fabrication Enter- prises, Inc: White Plains, New York) was used by the clinical staff before and after the patient's rehabilitation to document the initial and subsequent range of motion, evaluate their progress and to determine the level of disability. We used the goniometer, to assess the physical therapy effectiveness of the VR rehabilitation and to personalize the system's range of motion for each patient. We examined the differences between a range of movements limb join (flexion, extension, abduction, and adduction) before and after the VR rehabilitation. The greater the range of movement the better.
Paediatric Quality of Life Inventory (PedsQL) (Version 4.0 - UK English) results | Three weeks
  PedsQL is a standardised assessment for children aged 5-18 and was completed by patients before and after the IVR rehabilitation at-home trial. The scale features twenty-three items representing five dimensions: Physical, Emotional, Social, and School Functioning (e.g., physical functioning (problems with...) walking 100 metres; emotional functioning (problems with...) feeling afraid or scared; social functioning (problems with...) getting along with other children; and school functioning (problems with...) paying attention in class). The instructions ask how much of a problem each item has been in the past month, and responses are on a five-point scale ranging from 0 (never a problem) to 4 (almost always a problem) (Upton et al., 2005).
System Usability Scale (SUS) results | Three weeks
  System Usability Scale SUS) is a quantitative scale to measure system usability was completed by patients after the IVR rehabilitation at-home trial. It consists of a 10 item with 5-point response options from Strongly agree to Strongly disagree (Brooke, 1996). The scale evaluates the perceived ease of use (a single dimension). However, recent research shows that items 4 and 10 could provide the learnability dimension. Score contribution of each item was coded from 0 to 4 (items with positive words 1, 3, 5, 7 and 9; items with negative words 2, 4, 6, 8 and 10), and the sum of the contributions of the item scores was multiplied by 2.5 to obtain the overall SUS score (0 to 100). Scores were analysed above or below the standard mean score of 68. A score close to 100 was considered good usability of the system.
Interview Qualitative Results, Perceptions, Usability and Effectiveness of IVR system in ULMI rehab in children at home | Three weeks
  Semi-structured interviews were conducted by the research nurse in person (Pt 1, 4, 6, 7) and by phone (Pt 2, 3, 8) with patients and parents after the IVR rehabilitation at-home trial. Open-ended questions provided qualitative data relating to difficulty, pain and enjoyability, and participant attitudes towards the IVR system and its future deployment. Another semi-structured interview was conducted with the OT by the research nurse in person at the end of the trial to explore her attitudes towards the IVR system and future VR deployment. Both interviews were recorded, transcribed and anonymised.
Interview Quantitative Results, Perceptions, Usability and Effectiveness of IVR system in ULMI rehab in children at home | Three weeks
  During the semi-structured interview four ad-hoc closed ten-point Likert questions were asked. These provided a quantitative measure of the perceived ease or difficulty of use, pain levels and enjoyability of the IVR system.

CONTACTS AND LOCATIONS:
Locations (1):
- Ivan Phelan, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phelan I, Carrion-Plaza A, Furness PJ, Dimitri P. Home-based immersive virtual reality physical rehabilitation in paediatric patients for upper limb motor impairment: a feasibility study. Virtual Real. 2023 Jan 14;27(4):1-16. doi: 10.1007/s10055-023-00747-6. Online ahead of print. PMID 36686613